CLINICAL TRIAL: NCT03018431
Title: Impact of CT Scan and Lung Ultrasonogrpahy in Early Diagnostic Accuracy for Ventilation Acquired Lower Respiratory Tract Infections in Intensive Care Units.
Brief Title: CT Scan and Lung Ultrasonography to Improve Diagnostic of Ventilation Acquired Pneumonia in ICU
Acronym: ECTOPICUS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Principal Investigator, Paul-Henri WICKY, Medicla Doctor, Centre Hospitalier Universitaire de Besancon
Other Study IDs: CHBesançon
Record Dates: First submitted 2017-01-10; First posted 2017-01-12 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Ventilator-Associated Pneumonia; Tracheobronchitis
Keywords: Lung ultrasonography; Chest CT scan; ventilator-associated pneumonia; ventilator-associated tracheobronchitis; antibiotic stewardship
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Physician routine evaluation: systematic evaluation of the probability of tracheobronchitis or pneumonia based upon clinical and biological, associated with standard radiographs, performed by the physician in chrage of the patient.
- independent evaluation: systematic evaluation of the probability of tracheobronchitis or pneumonia based upon early CT scan, and repeated lung ultrasonography, performed by an independent operator.
  Interventions: Other: CT Scan

INTERVENTIONS:
Other: CT Scan — patients undergoing chest CT scan at admission and repeated lung ultrasonography
  Other Names: Ultrasonography
  Groups: independent evaluation

SUMMARY:
We aim to show that systematic ultrasonography performed in ventilated patients suspected of ventilation-acquired pneumonia could improve the accuracy of diagnostic of pneumonia, and helps defining the diagnostic of tracheobronchitis when lower respiratory tract infection is considered.

Chest CT scan is often performed before or just after admission in ICU, and usually show abnormalities that are revealed later on standard radiographs.

This last exam is traditionally considered as the gold standard to prove new pulmonary infiltrates, but the correlation with parenchymal consolidation is pretty low, and lead to over-diagnosing pneumonia, thus leading to a massive and maybe sometimes unconsidered prescription of antibiotic therapy.

Lung ultrasonography conducted systematically within the 3 first days after suspcion of pneumonia could help making the difference between real infection-linked lesions, and banal abnormalities following the hydric inflation of intra-thoracic organs, for instance pulmonary edema or pleural effusion.

An independent evaluation using lung ultrasound, and analysis of CT scan acquisition when performed, compared with the physician in charge of the patient appreciation by suggesting him to provide his own probability of pneumonia upon routine clinical and biological datas.

DETAILED DESCRIPTION:
Diagnostic of VAP and tracheobronchitis is often difficult in UC under mechanical ventilation, and usually occuring quite early after initial phase of hemodynamic instability, and characterized by needs of massive fluids supports and drugs infusion. The goldstandard is still standard chest X-ray, providing a picture of the whole abnormalities due to cardiac failure, and cardiogenic pulmonary edema. The high rate of water in chest of the patients under ventilation assistance and hemodynamic support is responsible of a misinterpretation of the abnormalities visualized on the radiographs. It is often considered that Lung ultrasonography is useful to appreciate the involvement of pleural effusion, explaning etiologies of hypoxemia, where cardiac failure is excluded by the simultaneous ultrasonographic evaluation. However, it is not well recognized that pulmonary parenchyma can be explored through echography, and that it provides a lot of information about the amount of liquid inside it, and the default of aeration. Thus, it can in real time help the physician to guide the therapeutics and manage the ventilation better. Moreover, the suspicion of infection, clinically and biologically leads to the early prescription of antibiotics, given that the radiography is abnormal. Knowing that there is now parenchymal consolidation but rather effusion or a certain degree of pulmonary edema could help avoiding treating falsely a respiratory infection.

The same thoughts can be held concerning Chest CT Scan, an exam often realized at the early stage of management in a critical situation. We can take for granted that when occurring in the 48 first hours of resuscitation, this exam shows in a certain number of cases preexisting abnormalities, that are revealed severla hours later by Chest radiograph, when the suspicion of respiratory infection acquired under ventilation emerge. If we take into account that these abnormalities seen on radiographs are just correlated to those that could be seen on CT, but with a certain delay, and are not de novo, it could lead to an overestimating of ventilation acquired pneumonia, because the criteria of a new radiographic infiltrate won't be valid anymore. The diagnostic of tracheobronchitis could then be more appropriated in a certain number of situations.

Our aim is to verify retrospectively by an adjudication committee, that this early CT Scan, within the 2 first days after admission if patient is ventilated and/or suspicion of lower respiratory tract infection, and a systematic lung ultrasonographic evaluation, provided by an independent operator, could change our appreciation of the frequency of ventilation-acquired pneumonia, comparing to the appreciation of th physician in charge of the patients.

We are thus conducting a repeated evaluation, at day 0, day 3 and day 7 with ultrasonography, in order to give a probability of pneumonia or tracheobronchitis by the echographist operator, and suggesting the physician to give his own probability based on clinical and biological routine datas. We then measure the rate of agreement between the two parts, to see how far the systematic evaluation using pleural ultrasonography could help defining the probability of infection, and validating the diagnostic of pneumonia. The impact should be to improve the accuracy within the first days 2 or 3 days after suspicion, when repeated, if possible by the same operator. One of the main benefit could be the reduction or better reevaluation of antibiotic therapy, if diagnostic of pneumonia is rejected secondary, eventually shorter course of treatment could be chosen, even if this point deserve to be evaluated in further studies.

ELIGIBILITY:
Inclusion Criteria:

* Immunocompetent subject,
* fever and/or purulent tracheal secretions and/or hyperleukocytosis or leukopenia, associated with a positive microbiological sample (within broncho-alveolar leakage, endotracheal aspiration, or distal sample),
* invasive mechanical ventilation initiated since at least 48hours, and suppose to be maintained for at least 48hours

Exclusion Criteria:

* Immunocompromised-patients defined by ; HIV treated or not, patient under corticotherapy, immunotherapy, inflammatory systemic diseases, solid organ transplant, solid tumor treated or not, bone marrow transplant or stem cells graft, hematological malignancy known or under treatment,
* moribond,
* ventilation expected to last less than 48hours,
* minor-aged patients,
* no social insurance or isolation,
* mental disability making the understanding of the purpose of too difficult.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every patient place under mechanical ventilation at least for 48 hours, suspected of lower respiratory tract infection, based on CDC criterias of ventilatior-acquired pneumonia.
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2017-10-15 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Concordance of diagnostic of tracheo-bronchitis or pneumonia under mechanical ventilation, between physician in charge and independent observator cunducting ultrasound and CT scan evaluation. | 8 days

SECONDARY OUTCOMES:
rate of agreement between radiographs, CT scan and lung ultrasonography | 8 days
correlation between evolution according to management of infection and misdiagnostic of pneumonia or tracheo-bronchitis or not by the clinician. | 8 days
  improving under treatment or worsening without antibiotic therapy when pneumonia diagnostic is valid or not, making further considering the management of antibiotic therapy by the physician guided by CT scan and/or ultrasonography.
  quantifying amount of situations when diagnostic of pneumonia is validated retrospectively by the adjudication, and delayed starting of antibiotics when diagnostic is not patent early in the standard evaluation, thus conducting to an increased risk of morbi-mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Lila Bouadma, MD,PhD, Study Director — Hôpital universitaire Bichat- Claude Bernard
Locations (2):
- France (2):
  - Hôpital Universitaire Jean Minjoz, Besançon, Doubs
  - Hôpital Bichat - Claude Bernard, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Haddam M, Zieleskiewicz L, Perbet S, Baldovini A, Guervilly C, Arbelot C, Noel A, Vigne C, Hammad E, Antonini F, Lehingue S, Peytel E, Lu Q, Bouhemad B, Golmard JL, Langeron O, Martin C, Muller L, Rouby JJ, Constantin JM, Papazian L, Leone M; CAR'Echo Collaborative Network; AzuRea Collaborative Network. Lung ultrasonography for assessment of oxygenation response to prone position ventilation in ARDS. Intensive Care Med. 2016 Oct;42(10):1546-1556. doi: 10.1007/s00134-016-4411-7. Epub 2016 Jun 20. PMID 27324241
- [Result] Mongodi S, Via G, Girard M, Rouquette I, Misset B, Braschi A, Mojoli F, Bouhemad B. Lung Ultrasound for Early Diagnosis of Ventilator-Associated Pneumonia. Chest. 2016 Apr;149(4):969-80. doi: 10.1016/j.chest.2015.12.012. Epub 2015 Dec 22. PMID 26836896
- [Result] Martin-Loeches I, Povoa P, Rodriguez A, Curcio D, Suarez D, Mira JP, Cordero ML, Lepecq R, Girault C, Candeias C, Seguin P, Paulino C, Messika J, Castro AG, Valles J, Coelho L, Rabello L, Lisboa T, Collins D, Torres A, Salluh J, Nseir S; TAVeM study. Incidence and prognosis of ventilator-associated tracheobronchitis (TAVeM): a multicentre, prospective, observational study. Lancet Respir Med. 2015 Nov;3(11):859-68. doi: 10.1016/S2213-2600(15)00326-4. Epub 2015 Oct 22. PMID 26472037
- [Result] Claessens YE, Debray MP, Tubach F, Brun AL, Rammaert B, Hausfater P, Naccache JM, Ray P, Choquet C, Carette MF, Mayaud C, Leport C, Duval X. Early Chest Computed Tomography Scan to Assist Diagnosis and Guide Treatment Decision for Suspected Community-acquired Pneumonia. Am J Respir Crit Care Med. 2015 Oct 15;192(8):974-82. doi: 10.1164/rccm.201501-0017OC. PMID 26168322